CLINICAL TRIAL: NCT06847815
Title: Determination of the Glycemic Index of Differently Processed Sweet Corn
Brief Title: Corn Glycemic Index
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB202500171; 2022-51181-38333 (Other Grant/Funding Number: US DEPT OF AG NATL INST OF FOOD AND AG)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Glycemic Index
Keywords: sweet corn; glycemic index

STUDY DESIGN:
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose Tolerance Drink (Active Comparator): 50 g glucose beverage
  Interventions: Other: Glucose Tolerance Drink
- Sweet corn (Experimental): Sweet corn providing 50 g of available carbohydrate
  Interventions: Other: Sweet corn

INTERVENTIONS:
Other: Sweet corn — Fresh and processed sweet corn
  Arms: Sweet corn
Other: Glucose Tolerance Drink — Beverage providing 50 g of glucose
  Arms: Glucose Tolerance Drink

SUMMARY:
Processing sweet corn may impact digestibility and, therefore, glycemic response following consumption. The primary aim of this study is to assess the glycemic index of various sweet corn products and varieties. An exploratory aim is to assess hunger/satiety scores following sweet corn intake.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent in English
* Willing to consume 50 g of glucose in less than 15 minutes (2 mornings)
* Willing to consume around 250 to 350 g of sweet corn in 10 to 15 minutes (3 mornings)
* Willing to provide 7 capillary blood samples by fingerstick (by fine lancet) during each 2-hour session

Exclusion Criteria:

* Metabolic disease or condition affecting blood glucose, such as diabetes type 1 and 2, metabolic syndrome, or polycystic ovary syndrome
* Baseline fasting blood glucose > 100 mg/dL
* Currently pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
iAUC | From enrollment to the end of 5 weeks.
  Incremental area under the glycemic response curve (iAUC)

SECONDARY OUTCOMES:
Hunger and Satiety Score | From enrollment to the end of 5 weeks.
  Hunger and Satiety Visual Analogue Scale from 0 to 100 mm (higher number indicates increased hunger, satisfaction, fullness, and eating perception)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Food Science and Human Nutrition Building, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided